CLINICAL TRIAL: NCT01059864
Title: Phase 2 Study Of The Effects Of Open-Label CP-690,550 And Double-Blind Atorvastatin On Lipids In Patients With Active Rheumatoid Arthritis
Brief Title: Study Of The Effects Of Atorvastatin On Cholesterol Levels In Rheumatoid Arthritis Patients Taking CP-690,550
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A3921109
Record Dates: First submitted 2010-01-28; First posted 2010-02-01 (Estimated); Results first posted 2012-12-13 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-11

CONDITIONS: Rheumatoid Arthritis
Keywords: cholesterol; lipids; rheumatoid arthritis; CP-690; 550
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tofacitinib; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: CP-690,550; Drug: Atorvastatin
- Arm 2 (Experimental)
  Interventions: Drug: CP-690,550; Drug: Atorvastatin Placebo

INTERVENTIONS:
Drug: CP-690,550 — 12 week open-label CP-690,550 10 mg oral tablets administered twice daily starting at Day 0 through Week 12
  Arms: Arm 1
Drug: Atorvastatin — Starting at Week 6 and continuing through Week 12 atorvastatin 10 mg oral tablets administered once daily
  Arms: Arm 1
Drug: CP-690,550 — 12 week open-label CP-690,550 10 mg oral tablets administered twice daily starting at Day 0 through Week 12
  Arms: Arm 2
Drug: Atorvastatin Placebo — Starting at Week 6 and continuing through Week 12 atorvastatin placebo tablets administered once daily
  Arms: Arm 2

SUMMARY:
All patients will be in instructed to eat a therapeutic lifestyle diet and will receive CP-690,550 throughout the 12 weeks of this study. After 6 weeks, half will receive the cholesterol lowering agent, atorvastatin, and half a matching placebo. This study will first measure the effects of CP-690,550 on cholesterol levels and then the effects of adding atorvastatin on those levels.

ELIGIBILITY:
Inclusion Criteria:

* must be diagnosed as having active rheumatoid arthritis
* agree to participate in the study and sign and informed consent document

Exclusion Criteria:

* History of serious infection within the past 6 months
* test positive for TB
* have any uncontrolled clinically significant disease or laboratory tests
* require administration of prohibited medications during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2010-02; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (11):
- United States (10):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Huntsville, Alabama
  - Pfizer Investigational Site, Gilbert, Arizona
  - Pfizer Investigational Site, Scottsdale, Arizona
  - Pfizer Investigational Site, Upland, California
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Dayton, Ohio
  - Pfizer Investigational Site, Mayfield Village, Ohio
  - Pfizer Investigational Site, Greenville, South Carolina
  - Pfizer Investigational Site, Allen, Texas
- Pfizer Investigational Site, Seoul, South Korea

REFERENCES:
- [Derived] Hetland ML, Strangfeld A, Bonfanti G, Soudis D, Deuring JJ, Edwards RA. Machine learning prediction and explanatory models of serious infections in patients with rheumatoid arthritis treated with tofacitinib. Arthritis Res Ther. 2024 Aug 27;26(1):153. doi: 10.1186/s13075-024-03376-9. PMID 39192350
- [Derived] Charles-Schoeman C, Hyde C, Guan S, Parikh N, Wang J, Shahbazian A, Stockert L, Andrews J. Relationship Between Paraoxonase-1 Genotype and Activity, and Major Adverse Cardiovascular Events and Malignancies in Patients With Rheumatoid Arthritis Receiving Tofacitinib. J Rheumatol. 2023 Jul 15:jrheum.2023-0112. doi: 10.3899/jrheum.2023-0112. Online ahead of print. PMID 37453736
- [Derived] Kristensen LE, Danese S, Yndestad A, Wang C, Nagy E, Modesto I, Rivas J, Benda B. Identification of two tofacitinib subpopulations with different relative risk versus TNF inhibitors: an analysis of the open label, randomised controlled study ORAL Surveillance. Ann Rheum Dis. 2023 Jul;82(7):901-910. doi: 10.1136/ard-2022-223715. Epub 2023 Mar 17. PMID 36931693
- [Derived] Hansen KE, Mortezavi M, Nagy E, Wang C, Connell CA, Radi Z, Litman HJ, Adami G, Rossini M. Fracture in clinical studies of tofacitinib in rheumatoid arthritis. Ther Adv Musculoskelet Dis. 2022 Dec 27;14:1759720X221142346. doi: 10.1177/1759720X221142346. eCollection 2022. PMID 36601090
- [Derived] Curtis JR, Yamaoka K, Chen YH, Bhatt DL, Gunay LM, Sugiyama N, Connell CA, Wang C, Wu J, Menon S, Vranic I, Gomez-Reino JJ. Malignancy risk with tofacitinib versus TNF inhibitors in rheumatoid arthritis: results from the open-label, randomised controlled ORAL Surveillance trial. Ann Rheum Dis. 2023 Mar;82(3):331-343. doi: 10.1136/ard-2022-222543. Epub 2022 Dec 5. PMID 36600185
- [Derived] Winthrop KL, Yndestad A, Henrohn D, Danese S, Marsal S, Galindo M, Woolcott JC, Jo H, Kwok K, Shapiro AB, Jones TV, Diehl A, Su C, Panes J, Cohen SB. Influenza Adverse Events in Patients with Rheumatoid Arthritis, Ulcerative Colitis, or Psoriatic Arthritis in the Tofacitinib Clinical Development Programs. Rheumatol Ther. 2023 Apr;10(2):357-373. doi: 10.1007/s40744-022-00507-z. Epub 2022 Dec 17. PMID 36526796
- [Derived] Winthrop KL, Curtis JR, Yamaoka K, Lee EB, Hirose T, Rivas JL, Kwok K, Burmester GR. Clinical Management of Herpes Zoster in Patients With Rheumatoid Arthritis or Psoriatic Arthritis Receiving Tofacitinib Treatment. Rheumatol Ther. 2022 Feb;9(1):243-263. doi: 10.1007/s40744-021-00390-0. Epub 2021 Dec 6. PMID 34870800
- [Derived] Cohen SB, Tanaka Y, Mariette X, Curtis JR, Lee EB, Nash P, Winthrop KL, Charles-Schoeman C, Wang L, Chen C, Kwok K, Biswas P, Shapiro A, Madsen A, Wollenhaupt J. Long-term safety of tofacitinib up to 9.5 years: a comprehensive integrated analysis of the rheumatoid arthritis clinical development programme. RMD Open. 2020 Oct;6(3):e001395. doi: 10.1136/rmdopen-2020-001395. PMID 33127856
- [Derived] Panaccione R, Isaacs JD, Chen LA, Wang W, Marren A, Kwok K, Wang L, Chan G, Su C. Characterization of Creatine Kinase Levels in Tofacitinib-Treated Patients with Ulcerative Colitis: Results from Clinical Trials. Dig Dis Sci. 2021 Aug;66(8):2732-2743. doi: 10.1007/s10620-020-06560-4. Epub 2020 Aug 20. PMID 32816215
- [Derived] Cohen SB, Tanaka Y, Mariette X, Curtis JR, Lee EB, Nash P, Winthrop KL, Charles-Schoeman C, Thirunavukkarasu K, DeMasi R, Geier J, Kwok K, Wang L, Riese R, Wollenhaupt J. Long-term safety of tofacitinib for the treatment of rheumatoid arthritis up to 8.5 years: integrated analysis of data from the global clinical trials. Ann Rheum Dis. 2017 Jul;76(7):1253-1262. doi: 10.1136/annrheumdis-2016-210457. Epub 2017 Jan 31. PMID 28143815
- [Derived] Cohen S, Radominski SC, Gomez-Reino JJ, Wang L, Krishnaswami S, Wood SP, Soma K, Nduaka CI, Kwok K, Valdez H, Benda B, Riese R. Analysis of infections and all-cause mortality in phase II, phase III, and long-term extension studies of tofacitinib in patients with rheumatoid arthritis. Arthritis Rheumatol. 2014 Nov;66(11):2924-37. doi: 10.1002/art.38779. PMID 25047021
- [Derived] McInnes IB, Kim HY, Lee SH, Mandel D, Song YW, Connell CA, Luo Z, Brosnan MJ, Zuckerman A, Zwillich SH, Bradley JD. Open-label tofacitinib and double-blind atorvastatin in rheumatoid arthritis patients: a randomised study. Ann Rheum Dis. 2014 Jan;73(1):124-31. doi: 10.1136/annrheumdis-2012-202442. Epub 2013 Mar 12. PMID 23482473
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921109&StudyName=Study%20Of%20The%20Effects%20Of%20Atorvastatin%20On%20Cholesterol%20Levels%20In%20Rheumatoid%20Arthritis%20Patients%20Taking%20CP-690%2C550

RESULTS

PARTICIPANT FLOW:
Groups:
- CP-690,550: Participants received CP-690,550 10 milligram (mg) tablet orally twice daily from Week 1 to 6 during open label run-in phase.
- CP-690,550 + Atorvastatin: Participants who received CP-690,550 10 mg tablet orally twice daily in open label run-in phase for 6 weeks were randomized to receive CP-690,550 10 mg tablet orally twice daily along with atorvastatin 10 mg tablet orally once daily from Week 6 to 12, during double-blind phase.
- CP-690,550 + Placebo: Participants who received CP-690,550 10 mg tablet orally twice daily in open label run-in phase for 6 weeks were randomized to receive CP-690,550 10 mg tablet orally twice daily along with placebo matched to atorvastatin 10 mg tablet orally once daily from Week 6 to 12, during double-blind phase.
Period: Open-Label Run-In Phase
Arm/Group | CP-690,550 | CP-690,550 + Atorvastatin | CP-690,550 + Placebo
Started | 111 | 0 | 0
Completed | 98 | 0 | 0
Not Completed | 13 | 0 | 0
Not completed — Adverse Event | 7 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0
Period: Double-Blind Treatment Phase
Arm/Group | CP-690,550 | CP-690,550 + Atorvastatin | CP-690,550 + Placebo
Started | 0 | 50 | 48
Treated | 0 | 50 | 47
Completed | 0 | 47 | 45
Not Completed | 0 | 3 | 3
Not completed — Adverse Event | 0 | 3 | 3

BASELINE CHARACTERISTICS:
Arm/Group | CP-690,550
Number analyzed (Participants) | 111
Age Continuous [Mean (Standard Deviation); unit: years] | 52.3 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline (Week 6) in Low Density Lipoprotein-Cholesterol (LDL-C) Level at Week 12
Time Frame: Baseline (Week 6), Week 12
Population: Full analysis set (FAS) included all participants who were randomized to the study treatment groups and received at least one dose of the randomized investigational drug (atorvastatin or placebo). Here 'N' (Number of Participants Analyzed) signifies those participants who were evaluable for this measure.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | CP-690,550 + Atorvastatin | CP-690,550 + Placebo
Number analyzed (Participants) | 46 | 45
percent change | -35.34 (2.25) | 5.80 (2.27)

2. Secondary Outcome: Change From Baseline in Low Density Lipoprotein-Cholesterol (LDL-C) at Week 12
Time Frame: Baseline (Week 6), Week 12
Population: FAS population included all participants who were randomized to the study treatment groups and received at least one dose of the randomized investigational drug (atorvastatin or placebo). Here 'N' (Number of Participants Analyzed) signifies those participants who were evaluable for this measure.
Measure: Least Squares Mean (Standard Error); unit: milligram per deciliter (mg/dL)
Arm/Group | CP-690,550 + Atorvastatin | CP-690,550 + Placebo
Number analyzed (Participants) | 46 | 45
milligram per deciliter (mg/dL) | -51.49 (2.99) | 5.30 (3.02)

3. Secondary Outcome: 12-Hours Fasting Lipid Profile
Description: Participants were required to fast for 12 hours prior to sampling for lipid profile which included following parameters: LDL-C, high-density lipoprotein-cholesterol (HDL-C), very low density lipoprotein-cholesterol (VLDL-C), total cholesterol, apolipoprotein A-1, apolipoprotein B, triglycerides (TGs) and Non-HDL-C.
Time Frame: Day 0, Week 2, 6 (Baseline), 10, 12
Population: FAS population included all participants who were randomized to the study treatment groups and received at least one dose of the randomized investigational drug (atorvastatin or placebo).
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | CP-690,550 + Atorvastatin | CP-690,550 + Placebo
Number analyzed (Participants) | 50 | 47
mg/dL
  Day 0: LDL-C | 111.99 (30.21) | 114.68 (30.54)
  Week 2: LDL-C | 124.87 (30.97) | 132.94 (34.90)
  Week 6 (Baseline): LDL-C | 135.83 (39.39) | 138.26 (39.07)
  Week 10: LDL-C | 80.58 (24.45) | 141.52 (35.17)
  Week 12: LDL-C | 84.03 (21.94) | 142.61 (35.72)
  Day 0: HDL-C | 54.96 (14.96) | 56.20 (14.18)
  Week 2: HDL-C | 61.11 (17.00) | 65.35 (15.12)
  Week 6 (Baseline): HDL-C | 67.39 (18.35) | 70.58 (18.00)
  Week 10: HDL-C | 70.12 (19.35) | 70.31 (18.42)
  Week 12: HDL-C | 71.09 (17.61) | 71.73 (16.40)
  Day 0: Total Cholesterol | 189.62 (39.26) | 196.58 (34.41)
  Week 2: Total Cholesterol | 213.11 (43.02) | 222.85 (40.50)
  Week 6 (Baseline): Total Cholesterol | 228.22 (47.93) | 234.27 (43.99)
  Week 10: Total Cholesterol | 174.42 (32.10) | 238.16 (40.18)
  Week 12: Total Cholesterol | 175.18 (29.24) | 240.49 (42.14)
  Day 0: Apolipoprotein A-1 | 139.48 (27.70) | 148.36 (26.25)
  Week 2: Apolipoprotein A-1 | 153.80 (31.11) | 168.13 (24.43)
  Week 6 (Baseline): Apolipoprotein A-1 | 164.18 (29.76) | 171.81 (28.02)
  Week 10: Apolipoprotein A-1 | 171.87 (30.47) | 172.30 (29.00)
  Week 12: Apolipoprotein A-1 | 171.02 (30.93) | 178.36 (28.55)
  Day 0: Apolipoprotein B | 90.30 (21.89) | 94.09 (20.04)
  Week 2: Apolipoprotein B | 96.18 (23.35) | 101.74 (22.78)
  Week 6 (Baseline): Apolipoprotein B | 100.28 (26.64) | 100.38 (22.05)
  Week 10: Apolipoprotein B | 69.32 (20.33) | 103.96 (23.63)
  Week 12: Apolipoprotein B | 70.35 (15.06) | 105.84 (23.48)
  Day 0: TGs | 113.54 (52.17) | 128.76 (69.17)
  Week 2: TGs | 135.69 (76.80) | 123.18 (62.51)
  Week 6 (Baseline): TGs | 127.16 (77.16) | 127.63 (58.48)
  Week 10: TGs | 117.90 (78.04) | 133.63 (84.23)
  Week 12: TGs | 100.78 (35.87) | 131.48 (56.66)
  Day 0: VLDL-C | 57.73 (49.23) | 70.41 (68.55)
  Week 2: VLDL-C | 81.48 (73.57) | 74.89 (65.42)
  Week 6 (Baseline): VLDL-C | 76.10 (71.63) | 75.30 (58.91)
  Week 10: VLDL-C | 69.00 (75.49) | 79.43 (66.86)
  Week 12: VLDL-C | 51.59 (33.38) | 78.64 (53.10)
  Day 0: Non-HDL-C | 134.66 (35.32) | 140.39 (33.75)
  Week 2: Non-HDL-C | 152.00 (39.84) | 157.50 (39.61)
  Week 6 (Baseline): Non-HDL-C | 160.83 (47.50) | 163.69 (41.96)
  Week 10: Non-HDL-C | 104.30 (32.65) | 167.85 (40.22)
  Week 12: Non-HDL-C | 104.09 (25.49) | 168.76 (39.90)

4. Secondary Outcome: 12-Hours Fasting Lipid Profile: Particle Size of Lipoproteins
Description: Participants were required to fast for 12 hours prior to sampling for lipid profile which included following parameters: plasma lipoprotein VLDL-C, LDL-C and HDL-C particles size.
Time Frame: Day 0, Week 2, 6 (Baseline), 10, 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: nanometer (nm)
Arm/Group | CP-690,550 + Atorvastatin | CP-690,550 + Placebo
Number analyzed (Participants) | 50 | 47
nanometer (nm)
  Day 0: VLDL-C Particles | 42.08 (6.68) | 46.15 (10.12)
  Week 2: VLDL-C Particles | 47.41 (11.86) | 47.31 (8.28)
  Week 6 (Baseline): VLDL-C Particles | 44.75 (6.41) | 48.67 (9.09)
  Week 10: VLDL-C Particles | 48.29 (8.65) | 47.48 (7.34)
  Week 12: VLDL-C Particles | 47.35 (7.40) | 47.58 (8.18)
  Day 0: LDL-C Particles | 21.19 (0.90) | 21.14 (0.74)
  Week 2: LDL-C Particles | 21.44 (0.77) | 21.55 (0.79)
  Week 6 (Baseline): LDL-C Particles | 21.65 (0.92) | 21.66 (0.81)
  Week 10: LDL-C Particles | 21.67 (0.86) | 21.45 (0.91)
  Week 12: LDL-C Particles | 21.74 (0.80) | 21.51 (0.80)
  Day 0: HDL-C Particles | 9.29 (0.44) | 9.21 (0.48)
  Week 2: HDL-C Particles | 9.25 (0.46) | 9.26 (0.48)
  Week 6 (Baseline): HDL-C Particles | 9.31 (0.50) | 9.30 (0.50)
  Week 10: HDL-C Particles | 9.33 (0.47) | 9.22 (0.53)
  Week 12: HDL-C Particles | 9.36 (0.45) | 9.25 (0.49)

5. Secondary Outcome: 12-Hours Fasting Lipid Profile: Level of Lipoprotein Particles
Description: Participants were required to fast for 12 hours prior to sampling for lipid profile which included following parameters: total and large VLDL-C and chylomicron particles (VLDLCP), medium and small VLDL-C particles; total, large, medium and small LDL-C particles; and intermediate density lipoprotein (IDL).
Time Frame: Day 0, Week 2, 6 (Baseline), 10, 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: nanomoles per liter (nmol/L)
Arm/Group | CP-690,550 + Atorvastatin | CP-690,550 + Placebo
Number analyzed (Participants) | 50 | 47
nanomoles per liter (nmol/L)
  Day 0: Total VLDLCP | 61.00 (38.88) | 56.20 (37.29)
  Week 2: Total VLDLCP | 68.89 (43.74) | 65.24 (41.56)
  Week 6(Baseline): Total VLDLCP | 73.23 (48.34) | 65.51 (41.39)
  Week 10: Total VLDLCP | 53.22 (42.36) | 70.07 (43.11)
  Week 12: Total VLDLCP | 45.07 (27.93) | 72.11 (37.22)
  Day 0: Large VLDLCP | 1.25 (2.14) | 2.79 (4.80)
  Week 2: Large VLDLCP | 3.09 (4.58) | 2.50 (3.63)
  Week 6(Baseline): Large VLDLCP | 2.43 (4.34) | 2.53 (3.63)
  Week 10: Large VLDLCP | 2.47 (4.57) | 2.85 (4.66)
  Week 12: Large VLDLCP | 1.45 (1.84) | 2.63 (3.48)
  Day 0: Medium VLDL-C Particles | 22.11 (22.14) | 23.26 (24.79)
  Week 2: Medium VLDL-C Particles | 27.20 (25.39) | 25.75 (27.62)
  Week 6 (Baseline): Medium VLDL-C Particles | 26.54 (23.72) | 24.59 (22.43)
  Week 10: Medium VLDL-C Particles | 25.36 (28.17) | 25.27 (21.74)
  Week 12: Medium VLDL-C Particles | 20.67 (12.95) | 25.46 (20.40)
  Day 0: Small VLDL-C Particles | 37.64 (19.93) | 30.15 (19.02)
  Week 2: Small VLDL-C Particles | 38.61 (20.27) | 36.98 (21.89)
  Week 6 (Baseline): Small VLDL-C Particles | 44.26 (27.94) | 38.39 (21.85)
  Week 10: Small VLDL-C Particles | 25.38 (18.80) | 41.94 (23.77)
  Week 12: Small VLDL-C Particles | 22.94 (17.39) | 44.01 (23.51)
  Day 0: Total LDL-C Particles | 1111.8 (336.45) | 1222.2 (350.51)
  Week 2: Total LDL-C Particles | 1175.9 (365.28) | 1201.7 (342.82)
  Week 6 (Baseline): Total LDL-C Particles | 1154.3 (440.45) | 1195.0 (352.53)
  Week 10: Total LDL-C Particles | 787.24 (282.87) | 1271.2 (381.29)
  Week 12: Total LDL-C Particles | 801.39 (285.35) | 1264.9 (410.30)
  Day 0: IDL Particles | 27.12 (31.90) | 30.98 (37.49)
  Week 2: IDL Particles | 36.58 (42.24) | 55.74 (55.78)
  Week 6 (Baseline): IDL Particles | 43.37 (52.14) | 53.94 (51.70)
  Week 10: IDL Particles | 24.46 (38.14) | 69.78 (74.08)
  Week 12: IDL Particles | 22.22 (39.47) | 66.91 (62.54)
  Day 0: Large LDL-C Particles | 451.88 (247.55) | 468.67 (191.87)
  Week 2: Large LDL-C Particles | 543.28 (225.96) | 589.28 (243.27)
  Week 6 (Baseline): Large LDL-C Particles | 581.73 (239.90) | 631.55 (266.98)
  Week 10: Large LDL-C Particles | 400.11 (175.75) | 582.04 (268.41)
  Week 12: Large LDL-C Particles | 424.26 (161.19) | 598.34 (241.53)
  Day 0: Total Small LDL-C Particles | 632.73 (401.86) | 722.46 (373.82)
  Week 2: Total Small LDL-C Particles | 596.12 (415.78) | 556.67 (399.91)
  Week 6 (Baseline): Total Small LDL-C Particles | 528.94 (501.32) | 509.45 (385.73)
  Week 10: Total Small LDL-C Particles | 362.72 (309.76) | 619.43 (445.00)
  Week 12: Total Small LDL-C Particles | 354.96 (313.20) | 599.77 (456.21)
  Day 0: Medium Small LDL-C Particles | 127.08 (83.27) | 149.43 (78.23)
  Week 2: Medium Small LDL-C Particles | 117.42 (83.36) | 114.74 (83.82)
  Week 6 (Baseline): Medium Small LDL-C Particles | 104.94 (99.40) | 108.19 (82.11)
  Week 10: Medium Small LDL-C Particles | 78.78 (64.95) | 130.57 (96.04)
  Week 12: Medium Small LDL-C Particles | 77.96 (66.36) | 124.20 (97.98)
  Day 0: Very Small LDL-C Particles | 505.59 (319.41) | 572.98 (296.63)
  Week 2: Very Small LDL-C Particles | 478.62 (333.47) | 441.93 (317.36)
  Week 6 (Baseline): Very Small LDL-C Particles | 424.02 (402.68) | 401.21 (305.54)
  Week 10: Very Small LDL-C Particles | 283.76 (246.26) | 489.00 (350.20)
  Week 12: Very Small LDL-C Particles | 276.93 (249.02) | 475.55 (359.14)

6. Secondary Outcome: 12-Hours Fasting Lipid Profile: Level of High Density Lipoprotein Cholesterol (HDL-C) Particles
Description: Participants were required to fast for 12 hours prior to sampling for lipid profile which included following parameters: total, large, medium and small HDL-C particles.
Time Frame: Day 0, Week 2, 6 (Baseline), 10, 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: micromole per liter (mcmol/L)
Arm/Group | CP-690,550 + Atorvastatin | CP-690,550 + Placebo
Number analyzed (Participants) | 50 | 47
micromole per liter (mcmol/L)
  Day 0: Total HDL-C Particles | 27.08 (5.74) | 29.58 (5.97)
  Week 2: Total HDL-C Particles | 30.89 (5.81) | 33.68 (5.74)
  Week 6 (Baseline): Total HDL-C Particles | 32.90 (5.94) | 35.44 (5.99)
  Week 10: Total HDL-C Particles | 34.57 (6.03) | 36.07 (6.89)
  Week 12: Total HDL-C Particles | 34.20 (5.63) | 35.77 (6.26)
  Day 0: Large HDL-C Particles | 8.88 (3.64) | 8.75 (4.13)
  Week 2: Large HDL-C Particles | 9.08 (4.17) | 9.56 (4.34)
  Week 6 (Baseline): Large HDL-C Particles | 10.04 (4.67) | 10.63 (4.69)
  Week 10: Large HDL-C Particles | 10.98 (4.39) | 9.93 (4.81)
  Week 12: Large HDL-C Particles | 11.23 (4.43) | 10.23 (4.34)
  Day 0: Medium HDL-C Particles | 3.74 (3.94) | 4.01 (3.63)
  Week 2: Medium HDL-C Particles | 3.87 (4.31) | 4.43 (4.41)
  Week 6 (Baseline): Medium HDL-C Particles | 3.89 (4.86) | 3.98 (3.90)
  Week 10: Medium HDL-C Particles | 4.57 (5.58) | 4.52 (4.12)
  Week 12: Medium HDL-C Particles | 3.85 (3.97) | 4.74 (4.59)
  Day 0: Small HDL-C Particles | 14.44 (6.15) | 16.80 (6.46)
  Week 2: Small HDL-C Particles | 17.94 (6.27) | 19.70 (6.83)
  Week 6 (Baseline): Small HDL-C Particles | 18.97 (6.35) | 20.83 (6.95)
  Week 10: Small HDL-C Particles | 19.04 (7.30) | 21.63 (6.17)
  Week 12: Small HDL-C Particles | 19.15 (6.19) | 20.79 (7.10)

7. Secondary Outcome: Disease Activity Score Using 28-Joint Count and C-Reactive Protein (3 Variables) (DAS28-3 [CRP])
Description: DAS28-3 (CRP) was calculated from the number of swollen joints (SJC) and painful joints (PJC) using the 28 joints count and the CRP (milligram per liter [mg/L]). DAS28-3 (CRP) less than or equal to (<=)3.2 indicated low disease activity, DAS28-3 (CRP) more than (>) 3.2 to 5.1 indicated moderate to high disease activity.
Time Frame: Day 0, Week 6 (Baseline), 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 + Atorvastatin | CP-690,550 + Placebo
Number analyzed (Participants) | 50 | 47
units on a scale
  Day 0 | 5.38 (1.24) | 5.23 (1.00)
  Week 6 (Baseline) | 3.44 (1.28) | 3.33 (1.10)
  Week 12 | 3.06 (1.26) | 2.99 (1.09)

8. Secondary Outcome: Disease Activity Score Using 28-Joint Count and C-Reactive Protein (4 Variables) (DAS28-4 [CRP])
Description: DAS28-4 (CRP) was calculated from the number of swollen joints (SJC) and painful joints (PJC) using the 28 joints count, C-reactive protein (CRP) [mg/L] and patient's global assessment (PtGA) of disease activity (participant rated arthritis activity assessment with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity). DAS28-4 [CRP] <=3.2 indicated low disease activity, DAS28-4 [CRP] >3.2 to 5.1 indicated moderate to high disease activity and DAS28 less than 2.6 indicates remission.
Time Frame: Day 0, Week 6 (Baseline), 12
Population: Since DAS28-3(CRP) and DAS28-4(ESR) are summarized, data for DAS28-4(CRP) was collected and reported in individual participant listings, but not statistically summarized for analysis as planned.
Arm/Group | CP-690,550 + Atorvastatin | CP-690,550 + Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Disease Activity Score Using 28-Joint Count and Erythrocyte Sedimentation Rate (3 Variables) (DAS28-3 [ESR])
Description: DAS28-3 (ESR) was calculated from the number of swollen joints (SJC) and painful joints (PJC) using the 28 joints count and the erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hr]). DAS28-3 (ESR) <=3.2 indicated low disease activity, DAS28-3 (ESR) >3.2 to 5.1 indicated moderate to high disease activity.
Time Frame: Day 0, Week 6 (Baseline), 12
Population: Since DAS28-3(CRP) and DAS28-4(ESR) are summarized, data for DAS28-3(ESR) was collected and reported in individual participant listings, but not statistically summarized for analysis as planned.
Arm/Group | CP-690,550 + Atorvastatin | CP-690,550 + Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Disease Activity Score Using 28-Joint Count and Erythrocyte Sedimentation Rate (4 Variables) (DAS28-4 [ESR])
Description: DAS28-4 (ESR) was calculated from the number of swollen joints (SJC) and painful joints (PJC) using the 28 joints count, the erythrocyte sedimentation rate (ESR) [mm/hr] and patient's global assessment (PtGA) of disease activity (participant rated arthritis activity assessment with transformed scores ranging from 0 to 10; higher scores indicated greater affectation due to disease activity). DAS28-4 (ESR) <=3.2 indicated low disease activity, DAS28-4 (ESR) >3.2 to 5.1 indicated moderate to high disease activity.
Time Frame: Day 0, Week 6 (Baseline), 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 + Atorvastatin | CP-690,550 + Placebo
Number analyzed (Participants) | 50 | 46
units on a scale
  Day 0 | 6.60 (1.32) | 6.44 (1.04)
  Week 6 (Baseline) | 4.33 (1.44) | 4.26 (1.15)
  Week 12 | 3.84 (1.57) | 3.81 (1.29)

11. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20) Response
Description: ACR20 responses were defined as greater than or equal to 20% improvement in tender or swollen joint counts and 20% improvement in 3 of the 5 remaining ACR-core set measures: 1) physician's global assessment of disease activity, 2) participants assessment of disease activity, 3) participants assessment of pain, 4) participants assessment of functional disability via a health assessment questionnaire, and 5) C-reactive protein at each visit.
Time Frame: Week 6 (Baseline), 12
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 + Atorvastatin | CP-690,550 + Placebo
Number analyzed (Participants) | 50 | 47
percentage of participants
  Week 6 (Baseline) | 76.0 | 76.6
  Week 12 | 82.6 | 65.2

12. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 50% (ACR50) Response
Description: ACR50 responses were defined as greater than or equal to 50% improvement in tender or swollen joint counts and 50% improvement in 3 of the 5 remaining ACR-core set measures: 1) physician's global assessment of disease activity, 2) participants assessment of disease activity, 3) participants assessment of pain, 4) participants assessment of functional disability via a health assessment questionnaire, and 5) C-reactive protein at each visit.
Time Frame: Week 6 (Baseline), 12
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 + Atorvastatin | CP-690,550 + Placebo
Number analyzed (Participants) | 50 | 47
percentage of participants
  Week 6 (Baseline) | 48.0 | 42.6
  Week 12 | 67.4 | 45.7

13. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70% (ACR70) Response
Description: ACR70 responses were defined as greater than or equal to 70% improvement in tender or swollen joint counts and 70% improvement in 3 of the 5 remaining ACR-core set measures: 1) physician's global assessment of disease activity, 2) participants assessment of disease activity, 3) participants assessment of pain, 4) participants assessment of functional disability via a health assessment questionnaire, and 5) C-reactive protein at each visit.
Time Frame: Week 6 (Baseline), 12
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 + Atorvastatin | CP-690,550 + Placebo
Number analyzed (Participants) | 50 | 47
percentage of participants
  Week 6 (Baseline) | 20.0 | 19.1
  Week 12 | 34.8 | 30.4

14. Secondary Outcome: Tender-Joint Count
Description: Tender joint count (TJC) is an assessment of 68 joints (upper body, upper extremity, and lower extremity). Each joint's response to pressure/motion was assessed using the following scale: Present/Absent/Not Done/Not Applicable (for artificial joints).
Time Frame: Day 0, Week 6 (Baseline), 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | CP-690,550 + Atorvastatin | CP-690,550 + Placebo
Number analyzed (Participants) | 50 | 47
tender joints
  Day 0 | 23.20 (18.15) | 21.38 (14.80)
  Week 6 (Baseline) | 10.48 (12.56) | 10.99 (13.22)
  Week 12 | 8.57 (12.83) | 7.83 (9.71)

15. Secondary Outcome: Swollen-Joint Count
Description: Swollen joint count (SJC): an assessment of 66 joints (upper body, upper extremity, and lower extremity). Each joint was assessed for swelling using the following scale: Present/Absent/Not Done/Not Applicable (for artificial joints).
Time Frame: Day 0, Week 6 (Baseline), Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | CP-690,550 + Atorvastatin | CP-690,550 + Placebo
Number analyzed (Participants) | 50 | 47
swollen joints
  Day 0 | 16.90 (12.67) | 15.34 (11.34)
  Week 6 (Baseline) | 6.36 (7.08) | 5.68 (5.94)
  Week 12 | 4.85 (5.51) | 5.15 (6.04)

16. Secondary Outcome: C-Reactive Protein (CRP)
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation. Normal range is 1-3 milligram per liter (mg/L).
Time Frame: Day 0, Week 6 (Baseline), 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | CP-690,550 + Atorvastatin | CP-690,550 + Placebo
Number analyzed (Participants) | 50 | 47
mg/L
  Day 0 | 33.17 (38.22) | 22.25 (26.96)
  Week 6 (Baseline) | 6.31 (11.76) | 3.34 (5.11)
  Week 12 | 6.04 (12.23) | 3.32 (5.23)

17. Secondary Outcome: Erythrocyte Sedimentation Rate (ESR)
Description: ESR is a laboratory test that provides a non-specific measure of inflammation. The test assesses the rate at which red blood cells fall in a test tube. Normal range is 0-30 mm/hr. A higher rate is consistent with inflammation.
Time Frame: Day 0, Week 6 (Baseline), 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | CP-690,550 + Atorvastatin | CP-690,550 + Placebo
Number analyzed (Participants) | 50 | 47
mm/hr
  Day 0 | 69.76 (36.40) | 60.32 (33.96)
  Week 6 (Baseline) | 37.42 (28.81) | 29.98 (20.46)
  Week 12 | 34.43 (27.02) | 30.31 (20.72)

18. Secondary Outcome: Patient Assessment of Arthritis Pain
Description: Participants assessed the severity of their arthritis pain using a 100 millimeter (mm) visual analog scale (VAS). The scale ranged from 0 (no pain) to 100 (most severe pain), measurement on a scale corresponds to the magnitude of their pain.
Time Frame: Day 0, Week 6 (Baseline), 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 + Atorvastatin | CP-690,550 + Placebo
Number analyzed (Participants) | 50 | 47
mm
  Day 0 | 65.66 (20.13) | 64.41 (27.40)
  Week 6 (Baseline) | 30.18 (21.91) | 31.26 (25.68)
  Week 12 | 25.72 (21.33) | 29.09 (25.11)

19. Secondary Outcome: Physician's Global Assessment (PhysGA) of Arthritis Pain
Description: The physician evaluated participants disease signs, functional capacity and physical examination independent of the patient's global assessment of arthritis. Physician's response was recorded using 0-100 mm visual analog scale (VAS), where 0=no pain and 100=most severe pain.
Time Frame: Day 0, Week 6 (Baseline), Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 + Atorvastatin | CP-690,550 + Placebo
Number analyzed (Participants) | 50 | 47
mm
  Day 0 | 63.28 (20.18) | 65.38 (24.86)
  Week 6 (Baseline) | 30.80 (22.09) | 31.85 (26.12)
  Week 12 | 24.30 (21.02) | 29.70 (25.17)

20. Secondary Outcome: Patient's Global Assessment (PtGA) of Arthritis Pain
Description: Participants answered: "Considering all the ways your arthritis affects you, how are you feeling today?" Participants responded by using a 0-100 mm visual analog scale where 0=no pain and 100=most severe pain.
Time Frame: Day 0, Week 6 (Baseline), Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | CP-690,550 + Atorvastatin | CP-690,550 + Placebo
Number analyzed (Participants) | 50 | 47
mm
  Day 0 | 68.10 (17.17) | 61.67 (18.72)
  Week 6 (Baseline) | 27.66 (18.03) | 28.08 (16.52)
  Week 12 | 23.33 (20.15) | 24.15 (15.91)

21. Secondary Outcome: Health Assessment Questionnaire Disability Index (HAQ-DI)
Description: HAQ-DI: participant-reported assessment of ability to perform tasks in 8 functional categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3, 0=least functional difficulty and 3=extreme functional difficulty.
Time Frame: Day 0, Week 6 (Baseline), 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 + Atorvastatin | CP-690,550 + Placebo
Number analyzed (Participants) | 50 | 47
units on a scale
  Day 0 | 1.54 (0.74) | 1.46 (0.74)
  Week 6 (Baseline) | 0.88 (0.71) | 0.88 (0.72)
  Week 12 | 0.74 (0.69) | 0.92 (0.78)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | CP-690,550 | CP-690,550 + Atorvastatin | CP-690,550 + Placebo
Serious Adverse Events (participants affected / at risk) | 2/111 | 0/50 | 1/47
Other Adverse Events (participants affected / at risk) | 15/111 | 21/50 | 19/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 (N=111) | CP-690,550 + Atorvastatin (N=50) | CP-690,550 + Placebo (N=47)
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 (N=111) | CP-690,550 + Atorvastatin (N=50) | CP-690,550 + Placebo (N=47)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Otorrhoea (Ear and labyrinth disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 1 | 0
Ocular vascular disorder (Eye disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 2 | 2
Pain (General disorders) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 5 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 2
Onychomycosis (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1
Tinea cruris (Infections and infestations) | 0 | 0 | 1
Tinea pedis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0
Blood potassium decreased (Investigations) | 0 | 1 | 0
Blood triglycerides increased (Investigations) | 0 | 1 | 0
Electrocardiogram abnormal (Investigations) | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 1
Weight increased (Investigations) | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Headache (Nervous system disorders) | 3 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1
Tinel's sign (Nervous system disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Sinus operation (Surgical and medical procedures) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.